CLINICAL TRIAL: NCT02013258
Title: Oxytocin Trial in Prader-Willi Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5208-N
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Prader Willi Syndrome
Keywords: Prader Willi syndrome; Oxytocin
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal oxytocin (Active Comparator): Intranasal oxytocin. 16 IU intranasal oxytocin x 5 days. One month interval between arms of treatment.
  Interventions: Drug: Intranasal oxytocin
- Placebo (Placebo Comparator): Placebo will be administered via nasal spray - 1 spray in each nostril x5 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Intranasal oxytocin — This is a double-blind placebo controlled 2x2 study. Subjects will receive OT for 5 consecutive days during their 7 day stay. This will be followed by a wash out period of 4-6 weeks.
  Other Names: Pitocin; Syntocinon
  Arms: Intranasal oxytocin
Other: Placebo — This is a double-blind placebo controlled 2x2 study. Placebo will be given via intranasal spray, one spray in each nostril daily x 5 days. One month interval between arms of treatment.
  Arms: Placebo

SUMMARY:
Individuals with Prader-Willi syndrome (PWS) have been found to have a deficit of oxytocin-producing neurons and decreased oxytocin receptor gene function, so the purpose of this study is to determine if oxytocin (OT) administration will improve some of the aspects of Prader-Willi syndrome that are particularly troublesome for children and their families (the insatiable appetite and social behaviors).

The research questions are:

1. Does intranasal oxytocin cause any side effects in children with PWS?
2. Does intranasal oxytocin administration alter appetite or behaviors in PWS?

DETAILED DESCRIPTION:
This study is to investigate if intranasal oxytocin will improve hyperphagia, social skills, and behaviors in subjects with Prader-Willi syndrome. This will be a randomized placebo controlled pilot study. The primary outcome measure is to determine if intranasal administration of oxytocin will cause any adverse events in subjects with Prader-Willi syndrome. Secondarily, the investigators will also perform evaluations to determine if intranasal oxytocin has any effect on social skills, behaviors, or appetite in children with Prader-Willi syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Children with genetically confirmed PWS
* Ages at ≥ 5 years and ≤ 11 years (must start treatment prior to 11th birthday)
* Child must be in nutritional phase 2b or 3, as determined by the PI at each site.
* Must currently be on growth hormone treatment, and have been receiving growth hormone treatment for at least one year prior to screening date.
* Treatment cannot have been interrupted for more than 1 week within 3 months prior to screening date.
* Priority will be given to children currently enrolled in the RDCRN Natural History study

Exclusion Criteria:

* Inability to tolerate intranasal administration of medication
* Hepatic insufficiency (AST/ALT greater than 3 times the normal levels for age)
* Renal insufficiency (BUN/Creatinine greater than 3 times the normal levels for age)
* History of an abnormal ECG (as determined by a cardiologist). If there is any question about cardiac function, ECG reports will be reviewed with a cardiologist prior to enrollment in the study.
* Child not receiving growth hormone treatment
* Child with hypertension or hypotension for age and sex (blood pressure >97% for age and sex or blood pressure <3% for age and sex)
* Diabetes mellitus
* Pregnant or lactating.
* Schizophrenia or psychosis
* Taking any psychotropic medications

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety of intranasal oxytocin in children with Prader-Willi syndrome | 3 months
  Occurrence of adverse event, description and quantification of clinical and behavior severity, pre- and post- intranasal oxytocin and placebo administration.

SECONDARY OUTCOMES:
Evaluation of food intake in Prader-Willi syndrome | 3 months
  Quantitative evaluation of hyperphagia via the Hyperphagia Questionnaire obtained on days 1, 4 and 6 during the 7 day study protocol and conducted in the evening on these days. Score will range from 0 (no hyperphagia behaviors) to 96 (most severe hyperphagia behaviors). Additionally quantity of food consumed will be recorded on Days 1,4, and 6.

OTHER OUTCOMES:
Evaluation of social effects of intranasal oxytocin in children with Prader-Willi syndrome | 3 months
  Evaluation of anxiety, food issues, irritability, social communication and behavioral issues will be measured on days 1, 4 and 6 using:
  1. Aberrant Behavior Checklist: Behavior rating scale used to measure behavior problems of children and adults with intellectual disabilities ages 6 - 54 years. Scores will range from 0 (no problem behaviors) to 174 (severe aberrant behaviors).
  2. Social Responsiveness Scale:designed to measure the breadth of repetitive behaviors. Scores will range from 64 (no repetitive behaviors) to 260 (severe repetitive behaviors).
  3. Repetitive Behavior Scales-Revised: Designed to measure the breadth of repetitive behaviors in autism spectrum disorder including: Ritualistic/Sameness Behavior; Stereotypic Behavior; Self-injurious Behavior; Compulsive Behavior; and Restricted Interests. Scores will range from 0 (no autistic behaviors) to 100 (severe autistic behaviors).
Effects of intranasal oxytocin on appetite-regulating hormones | 3 months
  Evaluation of plasma OT, ghrelin and other neuroendocrine hormones involved in appetite regulation (cortisol, orexin A, ghrelin, leptin, oxytocin, insulin).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Miller, MD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of California, Irvine, Orange, California
  - University of Florida, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas

REFERENCES:
- [Background] Tauber M, Mantoulan C, Copet P, Jauregui J, Demeer G, Diene G, Roge B, Laurier V, Ehlinger V, Arnaud C, Molinas C, Thuilleaux D. Oxytocin may be useful to increase trust in others and decrease disruptive behaviours in patients with Prader-Willi syndrome: a randomised placebo-controlled trial in 24 patients. Orphanet J Rare Dis. 2011 Jun 24;6:47. doi: 10.1186/1750-1172-6-47. PMID 21702900
- See also: Oxytocin treatment in children with Prader-Willi syndrome: A double-blind, placebo-controlled, crossover study. Miller JL, Tamura R, Butler MG, Kimonis V, Sulsona C, Gold JA, Driscoll DJ. Am J Med Genet A. 2017 May;173(5):1243-1250. — https://www.ncbi.nlm.nih.gov/pubmed/28371242